CLINICAL TRIAL: NCT06147349
Title: 2007 - Rene: Observational Study on the Occurrence of Possible Relapses and on the Quality of Life in Patients Who Underwent Radical Nefrectomy/Tumorectomy Surgery
Brief Title: Kidney Cancer Observational Protocol
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Montorsi, Professor, IRCCS San Raffaele
Other Study IDs: 2007 - Rene
Record Dates: First submitted 2023-10-10; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Renal Cancer
Keywords: Renal cancer; Radical Nephrectomy; Partial Nephrectomy; Relapse; Renal cancer diagnosis; Renal cancer treatment
MeSH Terms: conditions — Kidney Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients with kidney cancer who underwent radical or partial kidney removal surgery
  Interventions: Procedure: Radical or partial nephrectomy

INTERVENTIONS:
Procedure: Radical or partial nephrectomy — Removal of neoplastic mass either by full kidney excision or by targeted cancer removal

SUMMARY:
The aim of this observational study is to gather pre and post surgery clinical data belonging to patients who underwent radical or partial nephrectomy and to evaluate the impact of the surgery on the quality of life of the patients, as well as possible relapses within a 10 year period.

DETAILED DESCRIPTION:
A databasa was created with the intention of collecting data related to patients who underwent radical or partial nefrectomy surgery in an electronic case report form.

Each patient will be followed for 10 years approximately starting from the date of surgery for a total of 2 yearly visits for the first 5 years which could then be diluted in 1 visit per year for the remaining 5 years. At each visit control exams forseen by the standard care for post surgery patients will be evalued and tha data will then be transferred into the database. Yearly, a follow up questionnaire will be sent to the patients' home in order to obtain the information relative to possible relapses. The data collected will be handled following the most strict GCPs and privacy norms. The main objectives of the study are the collection and interpretation of the scientific data with the scope of: obtaining health benefits for the patients involved and for future patients with the same type of cancer, improving the scientific knowledge on the pathology and implementing new strategies for diagnosis and therapy and evaluating the epidemiologic changes of renal neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Kidney cancer diagnosis
* Indication to cancer removal through surgery
* Ability to read and sign the informed consent

Exclusion Criteria:

* Age < 18 years
* Absence of kidney cancer
* Inability to read and sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with kidney cancer who underwent radical or partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2010-01-27 (Actual); Primary Completion 2028-02-04 (Estimated); Study Completion 2028-02-04 (Estimated)

PRIMARY OUTCOMES:
Clinical parameter collection | 10 years
  Collection intended for the purpose of implementing diagnostic and therepautic strategies for the management of the disease in both the patient enrolled in the study and for future cases.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Montorsi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No